CLINICAL TRIAL: NCT04766502
Title: Study Evaluating the Bonds Between Circulating Tumoral ADN (ctDNA) and the Development of Peritoneal Carcinomatosis for Patients Treated With PIPAC
Brief Title: Bonds Between Circulating Tumoral ADN (ctDNA) and the Development of Peritoneal Carcinomatosis for Patients Under PIPAC
Acronym: PIPADN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2021-A00645-36
Record Dates: First submitted 2021-02-09; First posted 2021-02-23 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2024-12

CONDITIONS: Peritoneal Carcinomatosis
Keywords: PIPAC; Peritoneal Carcinomatosis; Circulating tumour DNA; Quality of Life
MeSH Terms: conditions — Peritoneal Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Blood sample (20ml) and Quality of Life Survey (Experimental)
  Interventions: Other: Blood sample (20 ml) and EORTC QLQC30 survey

INTERVENTIONS:
Other: Blood sample (20 ml) and EORTC QLQC30 survey — Blood sample (20ml) will be taken before and 24h after PIPAC procedure
  EORTC QLQC30 during pre operative consultation and at each post operative consultations

SUMMARY:
PIPADN is a pilot monocentric, study with a total duration of 42 months. The purpose of this study is to describe the variation of plasma ctDNA concentration between the 1st and the 3rd PIPAC session in patients with peritoneal carcinomatosis.

The improvement of life quality with this type of treatment will also be evaluated though the EORTC QLQ-C30 survey.

Each patient will have three PIPAC sessions spaced 6 to 8 weeks apart. Two blood samples will be taken during the first 3 PIPAC sessions, one the day before each procedure and a second one 24 hours afterwards.

The EORTC QLQ 30 survey will be completed by patients during the pre-operative consultation and at each post-operative consultation (about 3 weeks after PIPAC sessions).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* WHO 0 to 2
* Patient with cancer in the form of peritoneal carcinosmatois not eligible for cytoreduction surgery
* A histological diagnosis of the primary tumor or peritoneal carcinomatosis is essential.
* Patient with an indication for PIPAC for any reason (whether as part of a clinical research protocol or not). Patients with prior treatment with PIPAC are eligible.
* Patients with abdominal metastases or a single metastasis regardless of location (oligometastasis).
* For patients of childbearing age need for an effective method of contraception
* Informing patients and obtaining informed consent, dated and signed.
* Patient affiliated with a social security scheme

Exclusion Criteria:

* Age < 18 years old
* WHO > 3
* Patient who may benefit from cytoreduction surgery
* Patient with a contraindication to PIPAC
* Extra peritoneal disease with the exception of oligometastatic disease
* Persons deprived of liberty or under guardianship (including curatorship)
* Impossibility to undergo the medical follow-up of the trial for social, geographical or psychological reasons.
* For patients of childbearing age without an effective method of contraception
* Woman who is pregnant, likely to be pregnant, or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2025-01-07 (Actual)

PRIMARY OUTCOMES:
ctDNA | change from inclusion at 12 weeks
  ctDNA concentration change (ng/mL)
Peritoneal Regression Grading Score (PRGS) | at inclusion
  Results of each PIPAC will be evaluated using PRGS. PRGS (Peritoneal Regression Grading Score), going from 1 : no tumor cells, to 4 :solid growth in tumor cells
Peritoneal Regression Grading Score (PRGS) | an average of 6 weeks
  Results of each PIPAC will be evaluated using PRGS. PRGS : (Peritoneal Regression Grading Score), going from 1 : no tumor cells, to 4 :solid growth in tumor cells
Peritoneal Regression Grading Score (PRGS) | an average of 12 weeks
  Results of each PIPAC will be evaluated using PRGS. PRGS (Peritoneal Regression Grading Score), going from 1 : no tumor cells, to 4 :solid growth in tumor cells

SECONDARY OUTCOMES:
PIPAC discontinuation | an average of 6 week
  The reason (ei : progression, deterioration of the patient's general condition) of PIPAC discontinuation for patient who have had less than 3 PIPAC sessions
PIPAC discontinuation | an average of 12 weeks
  The reason (ei : progression, deterioration of the patient's general condition) of PIPAC discontinuation for patient who have had less than 3 PIPAC sessions
Peritoneal cancer index mesure | at inclusion
  Evaluation of disease extent
Peritoneal cancer index mesure | an average of 6 week
  Evaluation of disease extent
Peritoneal cancer index mesure | an average of 12 weeks
  Evaluation of disease extent
Quality of life mesure | At inclusion
  Quality of life will be mesured by EORTC Quality of Life C30 survey. EORTC : European Organization for Research and Treatment of Cancer. Measured from 0 to 35, 0 meaning minimal mictionnal discomfort, 35 meaning maximal mictionnal discomfort
Quality of life mesure | an average of 3 weeks
  Quality of life will be mesured by EORTC Quality of Life C30 survey. EORTC : European Organization for Research and Treatment of Cancer. Measured from 0 to 35, 0 meaning minimal mictionnal discomfort, 35 meaning maximal mictionnal discomfort
Quality of life mesure | an average of 9 weeks
  Quality of life will be mesured by EORTC Quality of Life C30 survey. EORTC : European Organization for Research and Treatment of Cancer. Measured from 0 to 35, 0 meaning minimal mictionnal discomfort, 35 meaning maximal mictionnal discomfort
Quality of life mesure | an average of 15 weeks
  Quality of life will be mesured by EORTC Quality of Life C30 survey. EORTC : European Organization for Research and Treatment of Cancer. Measured from 0 to 35, 0 meaning minimal mictionnal discomfort, 35 meaning maximal mictionnal discomfort

CONTACTS AND LOCATIONS:
Overall Officials: Cécilia CERIBELLI, MD, Principal Investigator — Institut de Cancérologie de Lorraine
Locations (1):
- Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No